CLINICAL TRIAL: NCT04917822
Title: Project KING: A Randomized Controlled Trial of Parallel Group Interventions to Strengthen Parent-child Relationship and Adaptation in Newly Arrived and Cross-boundary Families
Brief Title: Project KING: To Strengthen Parent-child Relationship and Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: International Social Services Hong Kong Branch (Unknown)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Project KING
Record Dates: First submitted 2021-04-12; First posted 2021-06-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Emotions; Family Conflict; Adaptation
Keywords: new immigrants; cross-boundary family; parallel group intervention

STUDY DESIGN:
Intervention Model Description: Both parents and children will be included in the intervention. The research team will conduct parallel intevention to parents and children in separate groups at the same time.
Who Masked: Participant
Masking Description: At the recruitment phase, the participants and the social workers who lead the intervention group will not know which intervention arm the participants will be assigned. A cluster of approximately 10 participants formed a group based on their attendance date in the intervention program. This group will be randomly assigned to one of the two intervention arms through pre-prepared randomization list calculated by random allocation software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion regulation arm (Experimental): The emotion regulation arm aims at improving emotional regulation skills among parents and children.
  Interventions: Behavioral: Emotion regulation
- Information provision arm (Active Comparator): The information provision arm aims at providing information about Hong Kong, such as education, community resources, medical care, employment, housing, and job-seeking among parents and children.
  Interventions: Behavioral: Information provision

INTERVENTIONS:
Behavioral: Emotion regulation — Emotion regulation arm will provide the parents and children with four 2-hour weekly sessions. For the parents, the main topics include raising awareness of emotions (e.g., learning emotions theories), developing skills to manage emotions (e.g., attention deployment, cognitive changes, response modification), and facilitating parent-child relationship (e.g., gratitude). For children, the main topics are similar to that in parents' intervention. In this arm, we give more specific examples and simple explanations to the children.
  Arms: Emotion regulation arm
Behavioral: Information provision — Information provision arm will provide the parents and children with four 2-hour weekly sessions. For the parents, the main topics in these four sessions include learning the general information about Hong Kong such as education and medical care, housing condition, employment and training. For children, the main topics include learning the general information about Hong Kong, such as education, community facility, and learning method.
  Arms: Information provision arm

SUMMARY:
This study aims at improving the emotional regulation strategies, enhancing the parent-child relationship and preventing family conflict among newly arrived and cross-boundary families in Hong Kong. We will provide one of the interventions to the participants: (a) the emotion regulation arm, which aimed at improving the emotion management skill for parent and child; or (b) the information provision arm, which aimed at providing information about Hong Kong, such as education, community resources, medical care, employment, housing, and job-seeking. We aim to recruit 200 parent-child pairs to participate in the study. The participants will be randomly assigned into an emotion regulation arm or an information provision arm. The ratio of the two arms is 3:2. Specifically, 120 and 80 parent-child pairs will be assigned to the emotion regulation arm and the information provision arm, respectively. The two intervention arms will provide four 2-hour weekly sessions to the participants. Before the intervention (T1), immediately after the intervention (T2), and one month after completing the intervention (T3), the participants will finish the assessments to evaluate the effectiveness of the intervention.

DETAILED DESCRIPTION:
1. Context of the study About 123 people migrate from Mainland China to Hong Kong to reunite with family every day. Migration from Mainland China to Hong Kong can be highly stressful. Newly arrived mothers and their children experience adaptation-related stressors, such as lifestyle changes, unhealthy housing conditions, and family financial restrictions, and they tend to experience high levels of psychological distress.

   Among the migrant population in Hong Kong, a particular group is known as cross-boundary children who engage in everyday-migration. Most cross-boundary children live in Shenzhen with their parents, who are not Hong Kong citizens. To attend school in Hong Kong, these children have to cross the border checkpoints connecting Hong Kong with mainland China every day. Families with cross-boundary children experience adaptation-related stressors, such as language difficulties, economic burden, and unclear citizenship status. These families have weaker social support networks in Shenzhen and seldom use community services in Hong Kong. Thus, cross-boundary families face multiple challenges and stressors due to their situation, which also puts them at a high risk of mental health problems.
2. Target of emotion regulation Newly arrived and cross-boundary families face similar problems, such as discrimination, acculturative stress, mental health problems (e.g., depression). All these problems can result in family conflict between parents and child. For example, early interviews have revealed that conflict over schoolwork and academic performance between children and parents could threaten overall family harmony. Frustrated with their lack of emotion regulation strategies, the children and parents often vented their anger and anxiety on each other, which sometimes led to physical abuse.

   Previous studies have demonstrated that the identification, comprehension, expression, regulation, and use of emotions are important predictors of individual adaptation and are positively correlated with mental health (e.g., happiness and social functioning). Parents' emotional regulation and mental health can influence their children's emotional socialization by means of diffusion through the family emotional climate. Thus, a community-based intervention focused on emotion regulation might help decrease these conflicts and enhance family harmony.
3. Cultural and contextual considerations in the intervention feature Family system theory states that families function as interdependent individual systems in which each member can impact others. It has been found that children's emotional problems are related to the stressful experiences and emotional symptoms of their parents. Therefore, we involved both parents and children concurrently in the intervention to maximize the intervention benefits. The parallel-group model is widely advocated in family-based intervention, but its implementation has a certain degree of difficulty. A parallel-group comprises two concurrent, but separate intervention groups (e.g., a child group together with a parent group); participants from the two groups engage in similar activities in different rooms with corresponding goals and contents. Compared with an intervention for individuals alone, involving family members in a family-based intervention can lead to greater benefits. Separating parents from children could prevent children from their parents' over-control and let each group deal with their own problems. The parallel-group model has been used to deal with different problems in parents and children. For example, a parent-child parallel-group helped improve the psychological functioning of depressed mothers, the mothers' caregivers, and children in Latino immigrant families. Therefore, the parent-child parallel group is considered an appropriate format for addressing the needs of cross-boundary families Two intervention studies evaluated the effectiveness of emotional regulation strategies on the parent-child relationship. The parental emotional management program increased emotional management strategy during the parent-child interaction, positive affect, subjective happiness, satisfaction with the parent-child relationship, and family harmony and decreased negative emotion among mothers of 6-8 years child in Hong Kong. However, this study did not include children in the intervention. A parent-child parallel emotional regulation group intervention improved the positive affect, resilience, and family harmony and reduced depressive symptoms among both parents and children. However, this study did not include the control group and had a small sample size.

   In sum, the present study aims to test the effectiveness of an emotion regulation parallel-group intervention on strengthening parent-child relationship and adaptation in newly arrived and cross-boundary families in Hong Kong.
4. Procedure We aim to recruit 200 parent-child pairs to participate in the study. The participants will be randomly assigned into one of the following arms: a) the relationship enhancement arm, which aims at improving emotional regulation skills among parent and child; b) the information provision arm, which aims at providing information about Hong Kong, such as education, community resources, medical care, employment, housing, and job-seeking. The ratio of the two arms is 3:2. Specifically, 120 and 80 parent-child pairs will be assigned to the relationship enhancement arm or the information provision arm, respectively. The two intervention arms will provide four 2-hour weekly sessions to the participants. The participants will finish the assessments at baseline (T1), immediately after the intervention (T2), and one month after completing the intervention (T3).

ELIGIBILITY:
For parents:

Inclusion Criteria:

1. came to Hong Kong for less than three years (newly arrived only);
2. provide care to at least one cross-boundary child (cross-boundary only);
3. have a child aged between 6-14
4. can participate in the group with the children at the same time;

Exclusion Criteria:

1. have a history of severe psychotic symptoms;
2. have previously participated in a similar intervention program.

For children:

Inclusion Criteria:

1. are 6-14 years of age;
2. have lived in mainland China for more than six months, and commuted daily between mainland China and Hong Kong (cross-boundary only);
3. have been studing in Hong Kong.

Exclusion Criteria:

1. have a history of severe psychotic symptoms;
2. have previously participated in a similar intervention program.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 217 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Emotional Management Strategy Questionnaire to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Emotional management strategy questionnaire is a 10-item scale assessing parents' and children's emotional management strategy. Possible scores range from 1 (not at all) to 6 (everyday). Higher scores indicate more frequent use of emotional management strategy.
Change from Baseline in Positive and Negative Affect Schedule to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Positive and negative affect schedule is a 10-item scale assessing parents' and children's positive and negative affect. Possible scores range from 1 (not at all) to 6 (everyday). Higher scores indicate more positive or negative affect.
Change from Baseline in Subjective Happiness Scale to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Subjective happiness scale is a 4-item scale assessing parents' and children's subjective happiness. Possible scores range from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate more subjective happiness.
Change from Baseline in Child-Parent Relationship Scale (Pianta) to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Child-parent relationship scale is a 4-item scale assessing the relationship between parents and children. Possible scores range from 1 (very dissatisfied) to 6 (very satisfied). Higher scores indicate better satisfaction with parents (or child).
Change from Baseline in Family Harmony Scale to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Family harmony scale is a 8-item scale assessing the family harmony. Possible scores range from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate better family harmony.
Change from Baseline in Adaptation Difficulties to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Adaptation difficulties is a 24-item scale assessing the adaptation difficulties after parents and children come to Hong Kong. Possible scores range from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate greater adaptation difficulties.
Change from Baseline in Self-developed Knowledge Questionnaire to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Knowledge questionnaire is a 18-item scale assessing how much parents and children know about Hong Kong (e.g., educaltional systems, community sevices). Possible scores include1 (right), 2 (wrong), and 3(don't know). Higher scores indicate greater knowledge about Hong Kong.

SECONDARY OUTCOMES:
Change from Baseline in Generalized Anxiety Disorder Questionnaire-7 to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Generalized anxiety disorder questionnaire assesses the anxiety symptoms among parents and children. Higher scores indicate more anxiety symptoms.
Change from Baseline in The Patient Health Questionnaire-9 to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Patient health questionnaire assesses the depressive symptoms among parents and children. Higher scores indicate more depressive symptoms.
Change from Baseline in Mental Health Inventory-5 to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Mental health inventory assesses the mental health among parents and children. Higher scores indicate better mental health.
Change from Baseline in 10-item Connor-Davidson Resilience Scale to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Connor-Davidson resilience scale assesses the individual resilience among parents and children. Higher scores indicate greater resilience.
Change from Baseline in Childhood Trauma Questionnaire to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Childhood trauma questionnaire whether parents spank their children. Higher scores indicate less physical abuse on children.
Change from Baseline in Child-Parent Relationship Scale (Driscoll & Pianta) to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Child-parent relationship scale has two subscales assessesing the closeness and conflict between parents and children, respectively. Higher scores indicate greater closeness or greater conflict between parents and children.
Change from Baseline in Self-Developed Service Use Questionnaire to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Self-developed service use questionnaire is a 14-item scale assessing whether parents and children use the social service in Hong Kong. Higher scores indicate more use of social service.
Change from Baseline in Self-Developed Capacity Questionnaire to Week 4 and to Week 8 | Baseline, week 4, and week 8
  Self-developed capacity questionnaire is a 11-item scale assessing whether parents and children have the capacity to use the social service in Hong Kong. Higher scores indicate greater capacity to use the social service.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy YU, Dr., Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data available to other researchers.

REFERENCES:
- [Background] Berwick DM, Murphy JM, Goldman PA, Ware JE Jr, Barsky AJ, Weinstein MC. Performance of a five-item mental health screening test. Med Care. 1991 Feb;29(2):169-76. doi: 10.1097/00005650-199102000-00008. PMID 1994148
- [Background] Brasseur S, Gregoire J, Bourdu R, Mikolajczak M. The Profile of Emotional Competence (PEC): development and validation of a self-reported measure that fits dimensions of emotional competence theory. PLoS One. 2013 May 6;8(5):e62635. doi: 10.1371/journal.pone.0062635. Print 2013. PMID 23671616
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Chan, A. K.-W., & Ngan, L. L.-S. (2018). Investigating the differential mobility experiences of Chinese cross-border students. Mobilities, 13(1), 142-156. https://doi.org/10.1080/17450101.2017.1300452
- [Background] Chan, K. L., Yeung, K. C., Chu, C. K., Tsang, K. Y., & Leung, Y. K. (2002). An evaluative study on the effectiveness of a parent-child parallel group model. Research on Social Work Practice, 12(4), 546-557. https://doi.org/10.1177/1049731502012004006
- [Background] Chan, P. W. K., & Kabir, A. H. (2014). Education across borders in Hong Kong. In H. Zhang, P. W. K. Chan, & C. Boyle (Eds.), Equality in education: Fairness and inclusion (pp. 155-166). Brill Sense. https://doi.org/10.1007/978-94-6209-692-9_12
- [Background] Dowell KA, Ogles BM. The effects of parent participation on child psychotherapy outcome: a meta-analytic review. J Clin Child Adolesc Psychol. 2010;39(2):151-62. doi: 10.1080/15374410903532585. PMID 20390807
- [Background] Driscoll, K., & Pianta, R. C. (2011). Mothers' and Fathers' Perceptions of Conflict and Closeness in Parent-Child Relationships during Early Childhood. Journal of Early Childhood & Infant Psychology.
- [Background] Fabrizio CS, Lam TH, Hirschmann MR, Pang I, Yu NX, Wang X, Stewart SM. Parental emotional management benefits family relationships: A randomized controlled trial in Hong Kong, China. Behav Res Ther. 2015 Aug;71:115-24. doi: 10.1016/j.brat.2015.05.011. Epub 2015 Jun 4. PMID 26112397
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lyubomirsky, S., & Lepper, H. S. (1999). A measure of subjective happiness: Preliminary reliability and construct validation. Social Indicators Research, 46(2), 137-155.
- [Background] Morris AS, Silk JS, Steinberg L, Myers SS, Robinson LR. The Role of the Family Context in the Development of Emotion Regulation. Soc Dev. 2007 May 1;16(2):361-388. doi: 10.1111/j.1467-9507.2007.00389.x. PMID 19756175
- [Background] Pianta, R. C. (1992). Child-parent relationship scale. Unpublished measure, University of Virginia, 11, 39-41.
- [Background] Qu D, Chen C, Kouros CD, Yu NX. Congruence and discrepancy in migrant children's and mothers' perceived discrimination: Using response surface analysis to examine the effects on psychological distress. Appl Psychol Health Well Being. 2021 Aug;13(3):602-619. doi: 10.1111/aphw.12249. Epub 2021 Feb 7. PMID 33554475
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Valdez CR, Padilla B, Moore SM, Magana S. Feasibility, acceptability, and preliminary outcomes of the Fortalezas Familiares intervention for latino families facing maternal depression. Fam Process. 2013 Sep;52(3):394-410. doi: 10.1111/famp.12033. Epub 2013 Jun 27. PMID 24033238
- [Background] Ward, C., & Kennedy, A. (1999). The measurement of sociocultural adaptation. International journal of intercultural relations, 23(4), 659-677. https://doi.org/10.1016/S0147-1767(99)00014-0
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] White, J. M., & Klein, D. M. (2002). Family theories. Sage.
- [Background] Xu, Y., Ann M. Farver, J., Zhang, Z., Zeng, Q., Yu, L., & Cai, B. (2005). Mainland Chinese parenting styles and parent-child interaction. International Journal of Behavioral Development, 29(6), 524-531. https://doi.org/10.1177/01650250500147121
- [Background] Yap MB, Allen NB, Sheeber L. Using an emotion regulation framework to understand the role of temperament and family processes in risk for adolescent depressive disorders. Clin Child Fam Psychol Rev. 2007 Jun;10(2):180-96. doi: 10.1007/s10567-006-0014-0. PMID 17265137
- [Background] Yu, N. X., Liu, I. K., & Bu, H. (2020). Enhancing resilience in cross-boundary families: A parent-child parallel group intervention. Journal of Social Work. https://doi.org/10.1177/1468017320919103
- [Background] Yu X, Stewart SM, Liu IK, Lam TH. Resilience and depressive symptoms in mainland Chinese immigrants to Hong Kong. Soc Psychiatry Psychiatr Epidemiol. 2014 Feb;49(2):241-9. doi: 10.1007/s00127-013-0733-8. Epub 2013 Jul 2. PMID 23818045
- [Background] Zhao, X., Zhang, Y., Longfei, L., & Zhou, Y. (2005). Evaluation on reliability and validity of Chinese version of childhood trauma questionnaire. Chinese Journal of Tissue Engineering Research, 9(16), 209-211.
- [Derived] Hu J, Bu H, Liu IKF, Yu NX. A Randomized Controlled Trial of Two Parent-Child Parallel Interventions to Enhance Positive Adaptation of Immigrant Families in Hong Kong: The Moderating Role of Depressive Symptoms. Behav Ther. 2024 Sep;55(5):1026-1042. doi: 10.1016/j.beth.2024.03.001. Epub 2024 Mar 20. PMID 39174263
- See also: Home Affairs Department and Immigration Department statistics on new arrivals from the Mainland (Fourth quarter of 2019). — https://www.had.gov.hk/file_manager/tc/documents/public_services/services_for_new_arrivals_from_the_mainland/report-2019q4.pdf
- See also: Home Affairs Department and Immigration Department statistics on new arrivals from the Mainland (First quarter of 2020). — https://www.had.gov.hk/file_manager/chs/documents/public_services/services_for_new_arrivals_from_the_mainland/report-2020q1_s.pdf